CLINICAL TRIAL: NCT07026682
Title: Comparison of Efficacy and Side Effect of Low Osmolar Oral Rehydration Solution Versus Oral Rehydration Solution For Malnourished Children (ReSoMal) in Management of Acute Watery Diarrhea in Severe Malnourished Children
Brief Title: Comparison of Low Osmolar ORS and ReSoMal for Treating Acute Watery Diarrhea in Severely Malnourished Children Aged 6 Months to 5 Years
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Sadaf Sumreen, Principal Investigator, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCHSLahore1
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Watery Diarrhea; Severe Acute Malnutrition in Childhood; Dehydration in Children
Keywords: Low Osmolar Oral Rehydration Solution; ReSoMal; Malnourished Children; Pediatric Diarrhea; Severe Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Low Osmolar ORS (Experimental): Received low osmolar oral rehydration solution (ORS) with an osmolarity of 245 mmol/L and sodium 75 mmol/L, administered orally according to WHO guidelines for rehydration in diarrhea.
  Interventions: Drug: Low Osmolar ORS
- Group ReSoMal (Active Comparator): Received ReSoMal oral rehydration solution specifically formulated for malnourished children, with lower sodium and higher potassium content, administered orally.
  Interventions: Drug: ReSoMal

INTERVENTIONS:
Drug: Low Osmolar ORS — Composition: Na⁺ 75 mmol/L, K⁺ 20 mmol/L, Cl- 65 mmol/L, citrate 10 mmol/L, glucose 75 mmol/L; osmolarity 245 mmol/L.
  Administered orally in rehydration regimen over 24 hours.
  Arms: Group Low Osmolar ORS
Drug: ReSoMal — Composition: Na⁺ 45 mmol/L, K⁺ 40 mmol/L, Cl- 76 mmol/L, citrate 7 mmol/L, glucose 125 mmol/L, Mg 6 mmol/L, Zn 300 µmol/L, Cu 45 µmol/L; osmolarity 300 mmol/L.
  Administered orally over 24 hours according to rehydration protocol.
  Arms: Group ReSoMal

SUMMARY:
Acute watery diarrhea is a common and serious health issue in children, especially in those who are severely malnourished. These children are at a much higher risk of complications such as dehydration, electrolyte imbalances, and even death. Oral Rehydration Solutions (ORS) are a widely used treatment to prevent and correct dehydration in such children. However, there are different types of ORS, and it is still unclear which one is more effective and safer for use in severely malnourished children.

This clinical study is being conducted at The Children's Hospital, Lahore, to compare two different types of ORS: low osmolar ORS and ReSoMal (a special rehydration solution designed for malnourished children). The aim is to determine which solution is more effective in correcting low potassium levels (a common problem in these children) and to identify which one has fewer side effects, particularly problems like low or high sodium levels that can be dangerous.

A total of 72 children between 6 months and 5 years of age, all diagnosed with severe malnutrition and mild to moderate dehydration due to acute watery diarrhea, will be included in the study. They will be randomly assigned to receive either low osmolar ORS or ReSoMal. Blood tests will be done before and after the treatment to check for changes in electrolyte levels. The frequency of diarrhea and the child's overall response to treatment will also be recorded.

The hypothesis of this study is that there is a significant difference in both effectiveness and side effects between the two ORS solutions. The results of this study will help doctors choose the safest and most effective ORS for treating diarrhea in severely malnourished children, improving care and potentially saving lives.

DETAILED DESCRIPTION:
After approval from ethical review committee of the hospital, 72 (36 in each group) severe malnourished children with watery diarrhea who present in the Department of Pediatrics Medicine University of Child Health Sciences,The Children's hospital Lahore will be included. Parents of the children who fulfill the above criteria will be counseled and explained the details of the study. Written informed consent and detailed history will be taken from each patient parent related to duration and frequency diarrhea. They will be divided into the following two groups using lottery method.

Group-I: Low osmolar ORS. (mmol/L: Na+ 75, K+ 20, Cl- 65, citrate 10, glucose 75, and osmolarity 245) Group-II: ReSoMal ORS. (Na 45 mmol/L, K 40 mmol/L, Cl 76 mmol/L, citrate 7 mmol/L, Mg 6 mmol/L, Zn 300 lmol/ L, Cu 45 lmol/L, glucose 125 mmol/L, osmolarity 300 mmol/L) At arrival in the hospital the dehydration status of the children will be assessed using the dehydration severity score (appendix). The weight of each child along with the height will be noted and I/V lines saved under aseptic measure. Base line investigations including the electrolytes and renal function tests will be sent to the lab and appropriate management of the infection with suitable antibiotics will be started. Fluid deficit will be corrected with 10 mL/kg/h of the assigned ORS given over the first 2 hours, then 5 mL/kg/h over a period of 10 to 12 hours until the deficit is corrected. Ongoing stool losses will be corrected with 5mL/kg after each watery or loose stool. The patients in group-I will receive low osmolar ORS fluid while the patients in group-II will receive standard ORS fluid. 24 hours after the fluid therapy started, blood will be drawn and will be sent for the measurement of electrolytes. The efficacy and side effects will be labelled as per operational definition. The frequency of passage of stool in the 24 hours will also be noted.

All data along will the lab values will be recorded into the attached performa, and all the labs will be done from the hospital lab.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 years.
* Both male and female.
* Children presenting with acute watery diarrhea.
* Children have mild to moderate dehydration.
* Children have serum sodium (135-145 mEq/L) and serum Potassium (2.5-3.4 mEq/L).
* Presence of severe malnutrition, defined as weight-for-length ≤ 3 standard deviations from the median of the World Health Organization (WHO) growth standards or mid-upper arm circumference (MUAC) <115 mm.
* Children tolerating oral fluid.
* Parent or guardian willing and able to provide informed consent for participation.

Exclusion Criteria:

* Critically ill children with shock, history of not passed urine for 6 h, convulsions and electrolyte abnormality requiring intravenous (IV) for severe dehydration.
* History of chronic gastrointestinal disorders, such as inflammatory bowel disease or celiac disease.
* Received antibiotics within 48 hours before enrollment.
* Children having any systemic illness requiring hospitalization or specific treatment, such as sepsis or pneumonia.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Correction of Hypokalemia After 24 Hours of Oral Rehydration | 24 hours after initiation of oral rehydration therapy
  This outcome assesses the proportion of participants whose serum potassium levels normalize after 24 hours of treatment with either low osmolar ORS or ReSoMal. Hypokalemia is defined as serum potassium <3.5 mmol/L. Correction is considered achieved if serum potassium rises to ≥3.5 mmol/L without requiring intravenous potassium supplementation.

SECONDARY OUTCOMES:
Incidence of Hyponatremia and Hypernatremia After 24 Hours of Oral Rehydration | 24 hours after initiation of oral rehydration therapy
  This outcome captures the number of participants who develop electrolyte imbalances, specifically hyponatremia (serum sodium <135 mEq/L) or hypernatremia (serum sodium >145 mEq/L), following 24 hours of rehydration with either low osmolar ORS or ReSoMal.

CONTACTS AND LOCATIONS:
Overall Officials: Sadaf Sumreen, Principal Investigator — University Of Child Health Sciences, Lahore
Locations (1):
- University Of Child Health Sciences, Lahore, Lahore, Punjab Province, Pakistan